CLINICAL TRIAL: NCT00665418
Title: Impact of High Concentrations of Sevoflurane on Laryngeal Reflex Responses in Pediatric Patients
Brief Title: Sevoflurane and Laryngeal Reflex Responses in Pediatric Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment finished earlier, because all 40 patients enrolled
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Albert Urwyler MD, Department of Anesthesia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNIBAS_UKBB_ANE_LR4; SNF_3200B0-109322
Record Dates: First submitted 2008-01-23; First posted 2008-04-23 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Laryngospasm
Keywords: Anesthesia; children; Larynx
MeSH Terms: conditions — Laryngismus; Laryngeal Diseases | interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: sevoflurane — sevoflurane 2.5% versus 4.7% (inhaled concentration) 10min each
  Other Names: Ultane

SUMMARY:
To describe laryngeal and respiratory reflex responses after controlled laryngeal stimulation in pediatric patients anesthetized with sevoflurane and to compare the evoked responses at two levels of anesthesia. To determine whether laryngeal and respiratory reflex responses after controlled laryngeal stimulation are completely suppressed in subjects when anesthetized with a MACEI95 (EI = endotracheal intubation) sevoflurane Hypothesis: The incidence of apnea with laryngospasm evoked by laryngeal stimulation will be reduced by 20% (from 25% to 5%) when the end-tidal concentration of sevoflurane is increased from 2.5% (MAC50) to 4.7% (MACEI95)

DETAILED DESCRIPTION:
Induction of anesthesia inhaling sevoflurane is a very common practice in pediatric anesthesia.However, unwarranted exaggerated upper airway defensive reflexes that develop into apnea and laryngospasm with resultant hypoxemia is more common and also more severe.

Despite their obvious clinical significance, reflexes that involve the function of the upper airway are only minimally understood and information on such reflexes is scarce in anesthetized humans. Nonetheless, a model was developed by analyzing respiratory variables and endoscopic images after stimulating the laryngeal mucosa with a small amount of distilled water. Clinical experience suggests that laryngeal reflexes occur more frequently under light levels of anesthesia. However, in contrast to other inhalational agents such as halothan, available data for sevoflurane suggest that an inverse correlation of laryngeal responsiveness to depth of hypnosis or end-tidal concentrations of sevoflurane (in adults and children) is less obvious. However, in all previous studies assessing laryngeal reflex responses under sevoflurane only low concentrations of sevoflurane (range of 1.0 - 2.5 Vol%) were examined. This is an important limitation because in clinical practice higher concentrations of sevoflurane are used, especially during manipulation of the airway, while the risk of airway irritation is high. Thus, the proposed study aims to explore the question whether the occurrence of laryngospasm can be reliably suppressed when high concentrations of sevoflurane are used.

Based on results of experiments assessing conditions that facilitate tracheal intubation, it is clear, that increasing the end-tidal concentration of volatile agents obtunds airway reflexes. Regarding intubation conditions, the concept of MACEI 50% or 95% describes the minimum alveolar concentration (MAC) of a volatile anesthetic needed by 50 or 95% of the patients, respectively, to prevent all movement during and immediately after tracheal intubation. The proposed study aims to assess respiratory reflex responses at these levels of anesthesia by analyzing the respiratory variables and endoscopic images. The incidences of well-defined airway reflexes (cough reflex, spasmodic panting, expiration reflex, and apnea with laryngospasm, central apnea) will be examined. Apnea with laryngospasm will be of primary interest in our study and digital video analysis of the glottic opening will allow for a detailed analysis of laryngeal performance.

ELIGIBILITY:
Inclusion Criteria:

* ASA I + II
* Elective intervention under general anesthesia

Exclusion Criteria:

* Reactive airway disease
* Respiratory tract infection (previous 2 weeks)
* Malignant hyperthermia
* Neuromuscular disease
* Cardiac disease

Ages: 25 Months to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Occurence of laryngospasm (defined as complete closure of the vocal or false cords with apnea lasting >10sec) after laryngeal stimulation | 5min

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O Erb, MD, Principal Investigator — Universitiy children's hospital Basel

REFERENCES:
- [Background] Oberer C, von Ungern-Sternberg BS, Frei FJ, Erb TO. Respiratory reflex responses of the larynx differ between sevoflurane and propofol in pediatric patients. Anesthesiology. 2005 Dec;103(6):1142-8. doi: 10.1097/00000542-200512000-00007. PMID 16306725